CLINICAL TRIAL: NCT00815165
Title: Cell-Mediated Immune Responses to Cytomegalovirus gB/MF59 Vaccine
Brief Title: Cytomegalovirus Cell-Mediated Immunity
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 06-0043; N01AI80007C
Record Dates: First submitted 2008-12-26; First posted 2008-12-29 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-09

CONDITIONS: Cytomegalovirus Infections
Keywords: cytomegalovirus, CMV, cell-mediated immunity, children, sub-study
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood.

GROUPS / COHORTS (2):
- Protocol 04-039 subjects: At least 50 and maximum of 100 healthy adolescent female subjects aged 12-17 years who were vaccinated in protocol 04-039 will be enrolled.
- Positive and Negative Controls: Approximately 100 screened subjects will be enrolled to serve as positive and negative controls.

SUMMARY:
Cytomegalovirus (CMV) is an important cause of illness and occasional deaths in infants who catch the virus before they are born, in newborns, and in children and adults who have weak immune systems. The purpose of this study is to look at how the CMV vaccine works in the blood. This study is being done along with the main CMV gB/MF59 vaccine study that looks at how the overall body reacts to the vaccine. Participants will include up to 100 healthy adolescent female subjects aged 12 to 17 years who were vaccinated in study 04-039 and 100 subjects that were screened for 04-039 to participate as controls. Study procedures will include up to 6 blood draws taken over a 13 month period. Participation will be about 31 months (unless the patient enrolls into the shedding study).

DETAILED DESCRIPTION:
Cytomegalovirus (CMV) is an important cause of morbidity and occasional mortality in congenitally infected infants and immuno-compromised children and adults, especially human immunodeficiency virus (HIV)-infected individuals and transplant recipients. Newborn infants represent a particularly high-risk group. This study of cell-mediated immune responses to cytomegalovirus GB/MF59 vaccine is a substudy of Division of Microbiology and Infectious Diseases, NIAID, NIH, DHHS (DMID) protocol 04-039, "A Randomized, Double-Blind, Placebo-Controlled, Phase II Study to Assess the Safety and Efficacy of the Cytomegalovirus gB/MF59 Vaccine in Preventing Systemic Cytomegalovirus Infection in Healthy Adolescent Females." This vaccine trial is designed to test the safety and efficacy of the CMV gB/MF59 vaccine. Primary goals of this study are to assess whether injection with 3 doses of the CMV gB/MF59 vaccine induces significant CD4+, CD8+ and/or regulatory T cell immune responses; to evaluate the boosting affect of gB/MF59 on the CMV-specific T cell responses after each of 3 doses of vaccine; to evaluate the persistence of CMV-specific T cell responses after vaccination; and to evaluate CMV-specific T cell responses in subjects that seroconvert during the vaccine trial. New techniques for the enumeration and characterization of antigen specific T cells are now available that will facilitate a precise analysis of the magnitude and functional capacity of influenza virus-specific T cells. All subjects enrolled in the CMV gB/MF59 trial at Vanderbilt and Cincinnati study sites will be eligible for enrollment in the cell-mediated immune response sub-study. Blood draws for assessment of cellular immune response will be obtained in 3 phases. Phase 1, N=50: at visit 1, the initial 100 consented subjects to recruit approximately 50 seropositive subjects (based on a 60 percent seropositive rate). Samples from this phase of the study will be used to establish the optimal conditions for the assay and to compare natural infection with vaccine induced T cell responses. Phase 2, N=50-100: at day 0 (before 1st dose of vaccine), day 30 (before the second dose of vaccine), day 60 (1 month after the second dose of vaccine), day 210 (1 month after the last dose of vaccine), and day 390 (7 months after the last dose of vaccine). Samples from this phase will be used to evaluate the boosting affect of gB/MF59 after each of 3 doses of vaccine and to evaluate the persistence of CMV-specific T cell responses. Phase 3: at each visit (S1-S8) for those subjects that seroconvert (i.e. if subject seroconverts at visit 10 blood will be obtained at visits S1-S8). These samples will be used to compare CMV-specific responses in subjects that either did or did not receive the vaccine and seroconvert during the study. These time points are based on the vaccine study design and the previous work evaluating T cell responses to vaccination 1 month and 6 months after immunization. Researchers will collect 30 ml of blood per draw in this trial enrolling up to 100 healthy adolescent females 12-17 years of age, inclusive. Blood volumes were determined to ensure sufficient numbers of cells to establish stimulation protocols and evaluate cell-mediated immune responses. The study duration will be 43 months. Subject duration will be 31 months, unless the subject seroconverts and enrolls into the shedding study. This study is linked to DMID protocol 04-039.

ELIGIBILITY:
Inclusion Criteria:

* Parent/legal guardian and subjects who understand and sign the assent as well as consent forms for this study.
* Subjects who qualify for the Division of Microbiology and Infectious Diseases, NIAID, NIH (DMID) study 04-039, "A Randomized, Double-Blind, Placebo-Controlled, Phase II Study to Assess the Safety and Efficacy of the Cytomegalovirus gB/MF59 Vaccine in Preventing Systemic Cytomegalovirus Infection in Healthy Adolescent," will be eligible for the initial pre-vaccination blood draw.
* Subjects who meet all inclusion criteria for the DMID 04-039 study and who are vaccinated will be allowed to participate in the remaining portions of this study.

Exclusion Criteria:

All subjects who are ineligible for the main DMID 04-039 study will not be eligible for the cell-mediated immunity sub-study.

Ages: 12 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A convenience sample of up to 100 healthy participants, ages 12-17 years, who were vaccinated in 04-039. Additionally, 100 screened subjects enrolled to serve as positive/negative controls.
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2006-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Immunogenicity based on cytomegalovirus (CMV) specific cell-mediated immunity. | Measured 30 days after the first dose, 30 days after the second dose, 30 days after the third dose and 7 months after the third dose of vaccine.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Cincinnati Children's Hospital Medical Center - Infectious Diseases, Cincinnati, Ohio
  - Vanderbilt University - Pediatric - Infectious Diseases, Nashville, Tennessee